CLINICAL TRIAL: NCT00949390
Title: Complementary and Alternative Medicine Usage Among Participants Enrolled in Phase I Oncology Clinical Trials
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0369
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Advanced Malignancy; Complementary and Alternative Medicine; CAM; Investigational Cancer Therapeutics; Phase I Clinical Trials
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Phase I and CAM Survey: Complementary and alternative medicine (CAM) in patients with advanced malignancies currently treated on University of Texas MD Anderson Cancer Center Phase I clinical trials.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Survey given at appointment time, then dropped in specified box anonymously.

SUMMARY:
Primary Objective:

· The primary objective is to estimate the prevalence of use of complementary and alternative medicine (CAM) in patients with advanced malignancies who are seen in the Phase I clinic at MD Anderson Cancer Center (MDACC).

Secondary Objective:

· Examine the association between prevalence of CAM use and demographic and socioeconomic characteristics (age, gender, race, income, and education level), participation in a phase I clinical trial, disease characteristics (diagnosis), patients' perceptions about their prognosis, physicians' information and permission for patients' CAM use, decision-making, and types of CAM used by patients.

DETAILED DESCRIPTION:
This survey study is intended to estimate the prevalence of use of CAM in patients who are currently being treated in the Phase I Clinical Trials Program at University of Texas MD Anderson Cancer Center. The survey includes questions about socioeconomic characteristics (age, gender, race, income, and education level), patients' diagnosis and patients' perceptions about their prognosis, physicians' information and permission for patients' use of CAM, patients' use of CAM (yes or no), decision-making (purpose of CAM use), resources and types of CAM.

Patients will be asked to drop the questionnaire into a box in a specified location after completion of the questionnaire. Accrual is expected to be 50-100 patients per month. This survey is expected to finish in 6 months.

ELIGIBILITY:
Inclusion Criteria:

1) Patients with a clinical diagnosis of malignancy who are seen in the outpatient oncology clinic.

Exclusion Criteria:

1) Presence of any clinically relevant condition that, in the opinion of the investigator/ coordinator, would interfere with completing the study including, but not limited to, visual problems, cognitive impairment or acute mental illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Current participation in a UT MDACC Phase I Clinical trial with a clinical diagnosis of advanced malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2009-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of CAM use among patients enrolled in Phase I clinical trials (Questionnaire Response Rate) | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org